CLINICAL TRIAL: NCT00256906
Title: Isolated Mild Fetal Ventriculomegaly and Neurodevelopmental Outcome
Status: Terminated | Type: Observational
Why Stopped: lack of funding
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Other Study IDs: IB1205-HMO-CTIL
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2007-06

CONDITIONS: Fetal Development
Keywords: lateral ventricles; fetal ventriculomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Isolated mild fetal ventriculomegaly is a common finding in fetal ultrasound examinations.

When the ventricular diameter is more than 15 mm it is usually considered as severe and connected to other malformations. Most of these children will be severely affected later in life. Less than 10 mm ventricular width considered as normal.

The current medical knowledge can not answer questions regarding future development of children who were diagnosed to suffer from mild (10-14.9 mm) brain ventriculomegaly during the pregnancy.

We would like to assess the development and neurological status of all children who were diagnosed as "mild ventriculomegaly" during the pregnancy in the last 6 years and to prospectively follow up all the children who will be diagnosed from the beginning of the study on for 6 years.

We hypothesized that the course of their development is different than of other children.

DETAILED DESCRIPTION:
Study design:

Patients:

1. All children who are currently 5-6 year-old who suffered from isolated fetal mild brain ventriculomegaly during the pregnancy.
2. All children who will be diagnosed with isolated fetal mild brain ventriculomegaly during the pregnancy from the beginning of the study for 6 years.

Methods:

1. All children will be examined by a pediatric neurologist who will perform a neuro-developmental assessment appropriate for age. The neurologist will decide individually whether there is a need for more medical tests.
2. All children will be assessed by a psychologist who will perform WIPPSI or BAYLEY tests according to age.

ELIGIBILITY:
Inclusion Criteria:

* All children who were or are diagnosed with isolated fetal mild ventriculomegaly

Exclusion Criteria:

* Anatomic malformations
* IVH
* Hydrocephalus
* Metabolic disorder
* CNS infection

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children up to the age of 10 years who were diagnosed with isolated mild ventriculomegaly as fetuses
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2006-01 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Itai Berger, MD, Principal Investigator — Hadassah University Medical Center
Locations (1):
- Itai Berger, Jerusalem, Israel